CLINICAL TRIAL: NCT01851603
Title: Phase I, Single-center, Inpatient, Randomized, Double-blind, Placebo-controlled, Dose Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles of Single Oral Doses of AVL-3288 (Anvylic-3288) Healthy Subjects.
Brief Title: Phase I Study to Evaluate the Safety and Pharmacokinetics of Oral Doses of Anvylic-3288 in Healthy Subjects
Acronym: AVL3288
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-1186; 1U01MH094247 (NIH)
Record Dates: First submitted 2013-05-06; First posted 2013-05-10 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVL-3288 (Experimental): Oral administration of AVL-3288
  Interventions: Device: AVL-3288
- Sugar pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: AVL-3288 — Drug
  Other Names: UCI-4083
  Arms: AVL-3288
Drug: Placebo — Identical diluent to that used for AVL-3288
  Other Names: Diluent solution
  Arms: Sugar pill

SUMMARY:
This is a brief inpatient study to determine the safety of a new drug in healthy people.

DETAILED DESCRIPTION:
AVL-3288, a "first in class" small molecule, selective allosteric modulator of the α7 nAChR, is implicated in the cognitive deficit in patients with neurologic and psychiatric disorders, including schizophrenia, Alzheimer's disease and attention deficit hyperactivity disorder. The mechanism of action, the allosteric modulation of α7 nAChR and improvement of cognitive and memory function both in relevant animal models and patients has been clearly described in recent literature. The effect of AVL-3288 strongly supports the rationale for use in schizophrenia given the dose effect relationship, peaking at a low dose in rats (HED 3 mg), in rodent schizophrenia and memory models. Phase I, single-center, inpatient, randomized, double-blind, placebo-controlled, dose escalating study to evaluate the safety, tolerability and pharmacokinetic profiles of single oral doses of AVL-3288 in healthy subjects. Subjects will be hospitalized in the University of Colorado Clinical Research Center (CTSA) for a 12 hour period after the single dose. Then there will be an ambulatory 24 and 48 hour observation and washout period of 10. Patients will receive an evoked potential measurement, the P50 sensory gating paradigm, and the Repeatable Battery for Assessment of Neuropsychological Status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Substance use. We do not accept inquiries by email.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 48 hours
  0,1,2,3, 4, 6, 8 ,12, 24, 48 hours post dose

SECONDARY OUTCOMES:
Number of participants with adverse events. | 10 days
  Corrected QT interval > 500 ms; hepatic enzyme > 3 times above the upper limit of normal values; systolic blood pressure > 200 mm Hg or diastolic blood pressure < 50 mm Hg.

OTHER OUTCOMES:
Repeatable Battery for Assessment of Neuropsychological Status Total Scale T Score | 24 hours
  T score on Total Scale of the Repeatable Battery for Assessment of Neuropsychological Status, differences between AVL-3288 or placebo arms and pretreatment baseline.
P50 Auditory Sensory Gating Ratio | 24 hours
  Ratio = (Conditioning P50 amplitude-Test P50 Amplitude)/Conditioning P50 Amplitude, differences between AVL-3288 or placebo arms from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — U of Colorado Denver
Locations (1):
- U of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Ng HJ, Whittemore ER, Tran MB, Hogenkamp DJ, Broide RS, Johnstone TB, Zheng L, Stevens KE, Gee KW. Nootropic alpha7 nicotinic receptor allosteric modulator derived from GABAA receptor modulators. Proc Natl Acad Sci U S A. 2007 May 8;104(19):8059-64. doi: 10.1073/pnas.0701321104. Epub 2007 Apr 30. PMID 17470817